CLINICAL TRIAL: NCT04928066
Title: Efficacy and Safety of Tofacitinib (TF) Combined With Iguratimod(IGU) in the Treatment of Moderate to Severe Active Rheumatoid Arthritis (RA)
Brief Title: The Efficacy and Safety of Tofacitinib (TF) With Iguratimod (IGU) on RA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Chief Physician, Qilu Hospital of Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tofacitinib-RA QiluH
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Tofacitinib; Iguratimod
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod; glucose utilization inhibitor; T 614; tofacitinib; prednylidene; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tofacitinib (TF)+Iguratimod (IGU) (Experimental): Drug: Iguratimod（IGU），25mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response.
  Drug: Tofacitinib（TF），5mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response.
  Drug: Prednisone （Pred）： 0-10mg, po, once per day (Qd) prescribed if needed and adjusted due to patient response.
  Interventions: Drug: Iguratimod; Drug: Tofacitinib; Drug: Pred
- Tofacitinib (TF) (Other): Drug: Tofacitinib（TF），5mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response.
  Drug: Prednisone （Pred）： 0-10mg, po, once per day (Qd) prescribed if needed and adjusted due to patient response.
  Interventions: Drug: Tofacitinib; Drug: Pred

INTERVENTIONS:
Drug: Iguratimod — Iguratimod tablet，25mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Other Names: IGU; T-614
  Arms: Tofacitinib (TF)+Iguratimod (IGU)
Drug: Tofacitinib — Tofacitinib,5mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Other Names: TF
Drug: Pred — Pred, 0-10mg, po, once per day (Qd) prescribed if needed and adjusted due to patient response.
  Other Names: Prednisone

SUMMARY:
RA is a common autoimmune disease that causes joint damage.It is necessary to reach the standard as soon as possible and give effective drugs according to the patient's disease activity to avoid disability. Tofacitinib(TF) is a new type of oral tyrosine kinase inhibitor (JAKi) for the treatment of moderate to severe active RA. However, there is alack of Chinese data on the joint scheme, long-term use, maintenance and stop of TF in the real world. We will use the new JAK combination regimen to treat RA patients, and carry out long-term clinical follow-up for 30 weeks.

DETAILED DESCRIPTION:
Objective: To observe the clinical efficacy and safety of TF combined with/ without IGU for 30 weeks in patients with moderate to severe active RA with different clinical characteristics and subgroups by using a prospective cohort , and to find the best combination scheme of TF.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following inclusion criteria will be eligible to participate in the study:

1. Patients who meet RA standards in 1987 and 2010 or ERA standards in 2012;
2. Age > 18 years old;
3. the extrapulmonary manifestations of RA were stable;
4. Patients with NSAIDs tolerance;
5. DAS28-ESR is highergreater than 2.6.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Patients with acute and chronic infection;
2. Platelet count < 80*10^9/L, or white blood cell < 3*10^9/L;
3. ALT or AST is 2 times higher than the upper limit of normal value;
4. Renal insufficiency: serum Cr ≥ 176 umol/L;
5. Pregnant or lactating women (breastfeeding);
6. Have a history of malignant tumor (the cure time is less than 5 years);
7. Patients with severe hypertension and cardiac insufficiency;
8. Other diseases or conditions in which immune suppressants cannot be used;
9. People who are allergic to TF.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who achieve clinical remission at week 30 using European League Against Rheumatism (EULAR) response criteria DAS28 | week 30
  The percentage of patients whose Disease Activity Score in 28 Joints (DAS28) achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2). The DAS28 is a composite score derived from 4 of these measures，that is the count of tender joint count（TJC, 0-28）and swollen joint count（SJC, 0-28）, measure erythrocyte sedimentation rate (ESR, mm/h) or C reactive protein (CRP, mg/L) and to make a patient assessment of disease activity i.e. 'global assessment of health' (GH) using a 100 mm visual analogue scale (VAS) with 0 = best, 100 = worst. DAS28 values were calculated as follows: DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x GH. High disease activity: DAS28-ESR > 5.1; Moderate disease activity: 5.1≥ DAS28 > 3.2 to 5.1; Low disease activity (LDA) and Remission mean Clinical remission.

SECONDARY OUTCOMES:
The percentage of patients who achieve clinical remission using DAS28-ESR at week 18 | week 18
  The percentage of patients whose DAS28 achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2) at week 18.
The percentage of patients who achieve clinical remission using DAS28-ESR at week 6 | week 6
  The percentage of patients whose DAS28 achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2) at week 18.
Percentage of Disease Activity Score 28 (DAS28) -ESR Criteria Responders at week 30 | week 30
  △DAS28 indicates the decline of DAS28-ESR from the baseline to week 30. EULAR response states were classified as follows: good responders were patients with an improvement from baseline (△DAS28-ESR) of > 1.2 and a DAS28-ESR at week 30 ≤ 3.2. Moderate responders: △DAS28 > 1.2 and still DAS28 > 3.2 at week 30, or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 30. Nonresponders：△DAS28 ≤0.6 or DAS28 >5.1 at week 30. DAS28-defined remission was classified as a score of <2.6.
Percentage of Disease Activity Score 28 (DAS28) -ESR Criteria Responders at week 18 | week 18
  EULAR response states were classified as follows: DAS28-ESR Good responders: △DAS28 > 1.2 and DAS28 ≤3.2 at week 18. Moderate responders：△DAS28 > 1.2 and still DAS28 > 3.2 at week 18; or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 18. Nonresponders：△DAS28 ≤0.6，or DAS28 >5.1 at week 18. DAS28-defined remission was classified as a score of <2.6.
Percentage of Disease Activity Score 28 (DAS28) -ESR Criteria Responders at week 6 | week 6
  EULAR response states were classified as follows: DAS28-ESR Good responders: △DAS28 > 1.2 and DAS28 ≤3.2 at week 6. Moderate responders：△DAS28 > 1.2 and still DAS28 > 3.2 at week 6; or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 6. Nonresponders：△DAS28 ≤0.6，or DAS28 >5.1 at week 6. DAS28-defined remission was classified as a score of <2.6.
Percentage of participants achieving ACR/EULAR remission at week 30 | week 30
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, Patient global assessment（PGA） ≤ 1 cm (on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease).
Percentage of participants achieving ACR/EULAR remission at week 18 | week 18
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, Patient global assessment（PGA） ≤ 1 cm (on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease).
Percentage of participants achieving ACR/EULAR remission at week 6 | week 6
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, Patient global assessment（PGA） ≤ 1 cm (on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease).
Change from baseline Simplified Disease Activity Index (SDAI) | up to week 30
  The SDAI is a composite score derived from these measures，that is the count of tender joint count（TJC, 0-28）, swollen joint count（SJC, 0-28）, C-reactive protein (CRP, mg/L), Patient global assessment（PGA）and physician global assessment（PHGA）, each of the last two was assessed on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease. SDAI score will be calculated with formula SDAI = TJC + SJC + PGA+PHGA+ CRP. SDAI score exceeding 26 is considered high disease activity; 11 <SDAI ≤26，moderate disease activity; 3.3 <SDAI ≤11, low disease activity; remission is SDAI score ≤ 3.3.
Change from baseline Clinical Disease Activity Index (CDAI) | up to week 30
  Change from baseline Clinical Disease Activity Index (CDAI) CDAI is a composite score derived from these measures，that is the count of tender joint count（TJC, 0-28）, swollen joint count（SJC, 0-28）, Patient global assessment（PGA）and physician global assessment（PHGA）, each of the last two was CDAI score will be calculated with formula CDAI = TJC + SJC + PGA + PHGA. CDAI > 22 is considered high disease activity; 10 <CDAI ≤ 22, moderate disease activity; 2.8 <CDAI ≤10, low disease activity; remission is CDAI score ≤2.8.
Change From Baseline in C-reactive Protein (CRP) | up to week 30
  Change from Baseline in C-reactive Protein (CRP), a component index of ACR20 and SDAI, CRP will be measured with blood samples.
Change From Baseline in Erythrocyte Sedimentation Rate (ESR) | up to week 30
  Change from Baseline in ESR, that is a component index of ACR20, DAS28-ESR and SDAI, ESR will be measured with blood samples.
Change from baseline Health Assessment Questionnaire Disability Index (HAQ-DI) | up to week 30
  Change from Baseline in HAQ-DI, a participant assessed measure of health assessment, shaveing eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item on a single scale has 4 degrees ranging from 0 (no functional difficulty) to 3 (unable to do), with higher scores indicating severe disease.
Percentage of American College of Rheumatology [ACR] 20 Criteria Responders every time | up to week 30
  Percentage of American College of Rheumatology [ACR] 20 Criteria Responders every time
Incidence of participant withdrawal | up to week 30
  Percentage of participants who withdraw from this study.
Number of participants with"adverse events (AEs)" | up to week 30
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with"adverse events (AEs)"i.e. physical exam abnormalities，vital sign abnormalities，laboratory value abnormalities，symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Yang, Dr., Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No